CLINICAL TRIAL: NCT07078916
Title: MOTOR TRAINING VERSUS MOTOR COGNITIVE TRAINING IN ATHLETES WITH CHRONIC ANKLE INSTABILITY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Jilan Adel yousef, lecturer of Physical Therapy for Musculoskeletal Disorders and its Surgeries, Faculty of Physical Therapy, kafrelsheikh University, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005726
Record Dates: First submitted 2025-07-14; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Chronic Ankle Instability, CAI
Keywords: Ankle Injuries [MeSH]; Ankle Sprain; Chronic Ankle Instability; Basketball Players; Balance Rehabilitation [MeSH]; Motor Skills [MeSH]; Cognitive Training [MeSH]; Visual Feedback; BlazePod; Dual-task Training; Dynamic Balance; Motor-Cognitive Training; Reaction Time
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Intervention Model Description: Double-blind parallel design randomized control study with allocation ratio 1:1
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor-Cognitive Training Group (OLBA + BlazePod™) (Experimental): Participants in this group will perform one-leg balance activities combined with visual feedback using BlazePod™
  Interventions: Behavioral: Motor-Cognitive Training Group (OLBA + BlazePod™)
- Motor Training Group (OLBA Only) (Active Comparator): Participants in this group will perform one-leg balance activities without any visual feedback.
  Interventions: Behavioral: Motor Training Group (OLBA Only)

INTERVENTIONS:
Behavioral: Motor-Cognitive Training Group (OLBA + BlazePod™) — Arm 1 participant will receive the One-leg-balance activity using visual feedback BlazePod technology as a dual motor-cognitive task training.
  Arms: Motor-Cognitive Training Group (OLBA + BlazePod™)
Behavioral: Motor Training Group (OLBA Only) — Arm 2 participant will receive a the One-leg-balance activity as a single motor task.
  Arms: Motor Training Group (OLBA Only)

SUMMARY:
This study aims to evaluate the effect of one-leg balance activity (OLBA) combined with visual feedback using BlazePod™ as a dual motor-cognitive rehabilitation task in basketball players with Chronic Ankle Instability (CAI). The intervention will be compared to OLBA alone as a motor task. Outcomes measured include dynamic balance, sense of instability, response time, athletic performance, and self-reported physical function. This study will help improve rehabilitation strategies for athletes suffering from ankle instability.

DETAILED DESCRIPTION:
* Chronic Ankle Instability (CAI) is a common condition among athletes, particularly basketball players, characterized by recurrent ankle sprains, impaired balance, and reduced functional performance. Effective rehabilitation strategies are crucial for restoring joint stability and preventing further injury.
* This study aims to compare the effects of motor-cognitive training versus motor training alone in basketball players with CAI. Participants will be randomly assigned into two groups: the first group will perform one-leg balance activity (OLBA) combined with visual feedback using BlazePod™ technology, while the second group will perform OLBA alone without visual feedback.
* The sample will be recruited from basketball teams through referral of athletes previously diagnosed with CAI, who continue to experience a feeling of ankle instability and recurrent "giving way" episodes at least one year after the initial lateral ankle sprain (LAS).
* The intervention will be conducted over 4 weeks, with 3 sessions per week. Each session will include 3 trials of the assigned OLBA task, with each trial lasting 30 seconds and a rest period of 1 minute between trials.
* The primary research question addressed by this study is: among basketball players with CAI, is there a significant difference between OLBA with visual feedback (BlazePod™) and OLBA alone in terms of dynamic balance, perceived instability, response time, athletic performance, and self-reported physical function?
* This study will contribute to the growing body of literature on dynamic balance training by comparing traditional motor tasks with dual-task training approaches that integrate cognitive-motor challenges using BlazePod™. BlazePod™ technology has demonstrated moderate to excellent reliability, particularly when used to provide feedback and monitor response during OLBA.
* Findings from this research may help healthcare professionals better understand the potential benefits of incorporating visual feedback and dual-task training into rehabilitation protocols for athletes with CAI. The results may also support the use of BlazePod™ as a tool for monitoring performance changes and facilitating motor learning in sports rehabilitation contexts.

ELIGIBILITY:
Inclusion Criteria:

* Young adult basketball athletes aged between (18 - 30) years.
* A history of unilateral one or more significant ankle inversion injury occurred at least 1 year before participation in the study.
* Interruption of physical activity or cessation from training for at least 24 hours following injury.
* Report episodes of giving way and sense of instability of the affected ankle.
* Two episodes of giving way or/ recurrent inversion injury should be reported by the patient before study enrollment at least two times in the last 6 months.
* Cumberland Ankle Instability Tool (CAIT) patient scores < 24.

Exclusion Criteria:

* A history of previous surgery or fracture to musculoskeletal structure (bone, joint, etc.) in the limb of the affected ankle.
* Acute lower limb sprain in the last 3 months before enrollment in the study resulting in interruption of physical activity for 1 day.
* Any disorder or disease that could affect the balance as vestibular disorders, eye injury, and so on.
* Any athlete who participates in any formal or informal rehabilitation.
* Participants who will not commit to two successive sessions will also be considered for exclusion.
* If they received NSAID 2 weeks before enrollment in the study.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Dynamic balance | At baseline and after 4 weeks of intervention
  Dynamic balance will be assessed using the Y-Balance Test, a reliable and valid tool for measuring postural control in three directions: anterior, posteromedial, and posterolateral.
  The participant will be asked to stand on the injured leg, then using another leg to reach the maximal point along the line in the three different directions, the directions named concerning the contact leg. The length of the line is normalized by the length of the patient's limb which is measured from ASIS to the medial malleolus.
  The goal of this test is to reach maximum excursion in every direction without shifting weight to or coming to rest on this foot of the reaching limb and then return the reaching limb to the beginning position in the center.
  Three trials in each direction to be familiarized. Actual trials will be 3 trials and best score will be calculated, The test will be conducted at baseline and after 4 weeks of intervention.
Sense of instability | The CAIT will be administered at baseline and after 4 weeks of intervention.
  Sense of ankle instability will be assessed using the Cumberland Ankle Instability Tool (CAIT), Consist of 32 points with a score less than 24 indicating CAI according to the International Ankle Consortium.
  The tool will be used in the Arabic version. The participants will be asked to choose the most suitable answer, with lower scores indicating greater perceived instability.
Response time. | Assessment will be conducted at baseline and after 4 weeks of intervention
  Response time will be measured through the BlazePod™ application, BlazePod™ is a method of motor learning assessment and cognitive motor training.
  BlazePod™ sensors are reactive lights that turn off or deactivate with contact, They are controlled via smartphone applications using Bluetooth low energy technology and allow for full customization of 10 colored lights which record time variables from activation until deactivation. In this scenario, pods will activate automatically and randomly with a timer and deactivate with the impact of the foot touching the top.
  Lower response time means better motor learning and is calculated automatically through the BlazePod application.
Self-reported physical function | The questionnaire will be administered at baseline and after 4 weeks of intervention.
  Self-reported physical function will be assessed using the Sport subscale of the Foot and Ankle Ability Measure (FAAM), a validated tool for evaluating functional limitations related to sports activities in individuals with foot and ankle disorders.
  The Sport subscale consists of 8 items, he response to each item on the Sports subscale is scored from 4 to 0, with 4 being "no difficulty" and 0 being "unable to do", scores on each item are added together to get the item score total, the highest potential score of the questioner is 32, The item score total is divided by the highest potential score.
  This value is multiplied by 100 to get a percentage, A higher score represents a higher level of physical function. with higher scores indicating better function.
  FAAM sport subscale will be used in Arabic version.

CONTACTS AND LOCATIONS:
Overall Officials: nasr awad abdelkader, Ph.D. in Physical Therapy, Principal Investigator — Assistant Professor of Physical Therapy for Musculoskeletal Disorders and its Surgeries, Faculty of Physical Therapy, Cairo University
Locations (1):
- Aman physical therapy center, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No